CLINICAL TRIAL: NCT00876226
Title: Study to Determine Steady-state Level of Citalopram Pharmacokinetic Parameters in Patients With Short Bowel Syndrome
Brief Title: Pharmacokinetics of Citalopram in Patients With Short Bowel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0479-07-FB
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Short Bowel Syndrome
Keywords: Citalopram; Pharmacokinetics; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacokinetics of Citalopram in Patients With Short Bowel Syndrome (Experimental): Citalopram pharmacokinetics will be studies in subjects with short bowel syndrome.
  Citalopram 20mg orally will be given to the subjects and on the seventh day blood will be drawn at hours 0,1,2,3,4,6,8,12,16 and 24 hours post-dose.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram — Citalopram pharmacokinetics will be studies in subjects with short bowel syndrome.
  Citalopram 20mg orally will be given to the subjects and on the seventh day blood will be drawn at hours 0,1,2,3,4,6,8,12,16 and 24 hours post-dose.
  Other Names: Celexa

SUMMARY:
This study will look at how the body interacts with citalopram in adult participants with short bowel syndrome. While information on depression in patients with short bowel syndrome is sparse, the investigators' experience is that these patients have a high incidence of depression and should benefit from a drug intervention.

DETAILED DESCRIPTION:
This prospective study will determine the pharmacokinetic parameters of citalopram in 12 adult patients with short bowel syndrome. While data on the prevalence of depression in patients with short bowel syndrome is sparse, the investigators' experience is that these patients have a high incidence of depression and should benefit from a psychopharmacological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages 19-65 years.
* Subjects must have less than 200cm of functional small intestine.
* Subjects must be at least one month post bowel resection.

Exclusion Criteria:

* Subjects less than 19 years or more than 65 years of age.
* Pregnant or breastfeeding women.
* Known hypersensitivity to citalopram or other SSRIs.
* Diagnosis of depression using MINI (Mini International Neuropsychiatric Interview).
* Ongoing antidepressant therapy.
* Evidence of cirrhosis (Child-Pugh stages B or C) or evidence of significant liver impairment defined as liver enzymes elevations greater that 2.5 times the upper limit of normal.
* Suicidal ideation.
* Bipolar disorder.
* Mania.
* Known history of seizures.
* Evidence of hyponatremia.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2012-09-11 (Actual); Study Completion 2012-09-11 (Actual)

PRIMARY OUTCOMES:
Measure plasma concentration of citalopram | Seven days
  Plasma concentration of citalopram (ng/mL) on the seventh day of treatment. Blood will be drawn at hours 0,1,2,3,4,6,8,12,16 and 24 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Sharma, MD, Principal Investigator — University of Nebraska

REFERENCES:
- [Background] Edes TE. Clinical management of short-bowel syndrome. Enhancing the patient's quality of life. Postgrad Med. 1990 Sep 15;88(4):91-5. doi: 10.1080/00325481.1990.11704755. PMID 2204906
- [Background] Cicalese L, Rastellini C, Sileri P, Abcarian H, Benedetti E. Segmental living related small bowel transplantation in adults. J Gastrointest Surg. 2001 Mar-Apr;5(2):168-72; discussion 173. doi: 10.1016/s1091-255x(01)80030-5. PMID 11331480
- [Background] Gulledge AD, Gipson WT, Steiger E, Hooley R, Srp F. Home parenteral nutrition for the short bowel syndrome. Psychological issues. Gen Hosp Psychiatry. 1980 Dec;2(4):271-81. doi: 10.1016/0163-8343(80)90080-8. PMID 6780408
- [Background] DiMartini A, Fitzgerald MG, Magill J, Funovitz M, Abu-Elmagd K, Furukawa H, Todo S. Psychiatric evaluations of small intestine transplantation patients. Gen Hosp Psychiatry. 1996 Nov;18(6 Suppl):25S-29S. doi: 10.1016/s0163-8343(96)00079-5. PMID 8937920
- [Background] Severijnen R, Bayat N, Bakker H, Tolboom J, Bongaerts G. Enteral drug absorption in patients with short small bowel : a review. Clin Pharmacokinet. 2004;43(14):951-62. doi: 10.2165/00003088-200443140-00001. PMID 15530127
- [Background] Broyles JE, Brown RO, Self TH, Frederick RC, Luther RW. Nortriptyline absorption in short bowel syndrome. JPEN J Parenter Enteral Nutr. 1990 May-Jun;14(3):326-7. doi: 10.1177/0148607190014003326. PMID 2112651
- [Background] Baumann P. Pharmacology and pharmacokinetics of citalopram and other SSRIs. Int Clin Psychopharmacol. 1996 Mar;11 Suppl 1:5-11. doi: 10.1097/00004850-199603001-00002. PMID 8732438
- [Background] Pollock BG. Citalopram: a comprehensive review. Expert Opin Pharmacother. 2001 Apr;2(4):681-98. doi: 10.1517/14656566.2.4.681. PMID 11336616
- [Background] Baumann P. Clinical pharmacokinetics of citalopram and other selective serotonergic reuptake inhibitors (SSRI). Int Clin Psychopharmacol. 1992 Jun;6 Suppl 5:13-20. PMID 1431018
- [Background] Milne RJ, Goa KL. Citalopram. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential in depressive illness. Drugs. 1991 Mar;41(3):450-77. doi: 10.2165/00003495-199141030-00008. PMID 1711447